CLINICAL TRIAL: NCT07090837
Title: Project Carer Matters 2: Evaluating the Effectiveness and Implementation of Caregiver Support Initiatives for Caregivers of Older Patients in Singapore
Brief Title: Evaluating the Effectiveness and Implementation of Caregiver Support Initiatives for Caregivers of Older Patients in Singapore
Acronym: PCM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Glass George Frederick Jr, Principal Investigator, Tan Tock Seng Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ECOS2024/00077
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Caregiver; Caregiver Stress; Caregiver Resilience and Stress
Keywords: Caregiver; Caregiver burden; Caregiver stress; Digital health; Caregiver support
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants receive the following interventions as deemed appropriate based on their caregiving and learning needs:
  1. CarePal: A one-stop resource library for caregivers of older adults
  2. Nasogastric tube (NGT) webapp: An electronic training platform to learn NGT feeding and management
  3. Carer OnBoard programme
  4. Caregiver resources in NHG Health App (NHA): Relevant healthcare professionals or TTSH staff will introduce caregivers to the resources they may need in the NHA app. ;
  5. Carer guide, a resource booklet providing information and community resources for caregivers.
  6. Group Caregiver Training, for caregivers who are able to attend group caregiver training (instead of learning at the bedside);
  7. NHG Care Telephonic team to provide telephonic support to caregivers post-discharge.
  8. Nurses or other healthcare professionals providing relevant information on community programmes
  Interventions: Other: Caregiver Support Model
- Control Arm (Placebo Comparator): Participants in this group will receive standard caregiver support
  Interventions: Other: Standard caregiver support

INTERVENTIONS:
Other: Caregiver Support Model — 1. CarePal: A one-stop resource library for caregivers of older adults
  2. Nasogastric tube (NGT) webapp: An electronic training platform to learn NGT feeding and management
  3. Carer OnBoard programme
  4. Caregiver resources in NHG Health App (NHA): Relevant healthcare professionals or TTSH staff will introduce caregivers to the resources they may need in the NHA app.
  5. Carer guide, a resource booklet providing information and community resources for caregivers.
  6. Group Caregiver Training, for caregivers who are able to attend group caregiver training (instead of learning at the bedside);
  7. NHG Care Telephonic team to provide telephonic support to caregivers post-discharge.
  8. Nurses or other healthcare professionals providing relevant information on community programmes
  Arms: Intervention arm
Other: Standard caregiver support — Participants are provided standard bedside caregiver education as appropriate and information reinforcement through leaflets and booklets
  Arms: Control Arm

SUMMARY:
We are evaluating the caregiver support initiatives at a tertiary hospital in Singapore (Tan Tock Seng Hospital - TTSH) provided to caregivers caring for older patients.

The evaluation will focus on 1) evaluating the process / delivery / implementation of these initiatives to caregivers and 2) the outcomes of caregivers and their care recipients after receiving these caregiver support services at TTSH. Research questions are as follows:

Process evaluation:

1. How are the bundle(s) of caregiver support initiatives at TTSH delivered to caregivers?
2. What and how was impact achieved for these initiatives?

   Outcome evaluation:
3. Did caregivers (and patients) benefit from these support initiatives and how?
4. Which aspects of the caregiver support initiatives are most beneficial to caregivers (and patients)?

Eligible caregivers will be invited to take part in the study and to complete 3 surveys and an optional interview over the period of their care recipients' hospital stay at TTSH, and 2 months after discharge. During their care recipients' stay, they may be introduced to any of the caregiver support initiatives, based on their needs. Caregivers enrolled in this study will take part in 3 surveys - 1 conducted at the beginning of care recipients' hospital stay, 1 conducted around the discharge period and 1 conducted one month after discharge. The aim of the surveys is to find out if caregivers have attended or used any of these services and whether they benefited from them.

DETAILED DESCRIPTION:
This is a mixed method study that seeks to evaluate the bundle of caregiver support initiatives being provided to caregivers at TTSH, based on their needs. The evaluation will focus on 1) evaluating the process / delivery / implementation of these initiatives to caregivers and 2) the outcomes of caregivers and their care recipients after receiving these caregiver support services at TTSH. Research questions are as follows:

Process evaluation:

1. How are the bundle(s) of caregiver support initiatives at TTSH delivered to caregivers?
2. What and how was impact achieved for these initiatives?

   Outcome evaluation:
3. Did caregivers (and patients) benefit from these support initiatives and how?
4. Which aspects of the caregiver support initiatives are most beneficial to caregivers (and patients)?

Quantitative methods:

Eligible caregivers will be invited to take part in the study and to complete 3 surveys and an optional interview over the period of their care recipients' hospital stay at TTSH, and 2 months after discharge. During their care recipients' stay, they may be introduced to any of the caregiver support initiatives, based on their needs. Caregivers enrolled in this study will take part in 3 surveys - 1 conducted at the beginning of care recipients' hospital stay, 1 conducted around the discharge period and 1 conducted one month after discharge. The aim of the surveys is to find out if caregivers have attended or used any of these services and whether they benefited from them.

We hypothesise that caregivers outcomes, for e.g. caregivers' knowledge, preparedness to provide care and well-being will be increased for those who have used or attended the initiatives recommended for them by the hospital and caregivers' stress, anxiety, depression, will decrease after receiving these caregiver support initiatives. We also hypothesise that the time spent on caregiving will decrease for those who have used or attended the hospital's caregiver support services and initiatives.

As some of the caregiver initiatives may be progressively implemented at TTSH over the study period, the study will capture data from caregivers who did not receive these initiatives with those who have received them when these initiatives were made available at the hospital.

We will also seek patients' consent to use their data in EPIC for research purposes. We hypothesise that patients' re-admission and visits to the ED post-discharge will be reduced.

Qualitative Methods:

Through the optional interviews with caregivers, either before or after discharge of the care recipients, we aim to ask the following research questions:

1. How were the caregiver support initiatives introduced and carried out at TTSH?
2. How did caregivers respond to these initiatives and what were their perceptions towards these interventions? Which aspects of these initiatives benefit them the most and why?
3. What are the barriers and facilitators faced by the healthcare professionals who implemented these initiatives to caregivers?

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and above
* Main or secondary caregiver of an older person receiving home-based care
* Able to read and converse in English
* Has a mobile smartphone and is able to navigate basic functionalities on mobile apps

Exclusion Criteria:

* Participants who are cognitively impaired
* Unwilling to download and utilise app
* Unable to read or converse in English comfortably

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Preparedness for Caregiving Scale | 1 month
  8-item scale measuring caregiver preparedness for caregiving. Average score ranges from 0 - 4, higher score indicating better preparedness for caregiving
Caregiver Resourcefulness Scale | 1 month
  8-item scale measuring caregiver resourcefulness. Total score calculated ranging from 8 - 40 with higher scores indicating higher resourcefulness
Zarit Burden Scale - 12 Item | 1 month
  12-item scale measuring caregiver burden. Total score calculated range from 0-48, with higher scores indicating higher burden

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 1 month
  14-item scale measuring anxiety and depression. Anxiety measured over 7 items, with score ranging from 0-21, with higher scores indicating higher anxiety. Depression measured over 7 items, with score ranging from 0-21, with higher scores indicating higher depression
EQ5D-5L | 1 month
  5-level EQ-5D version to measure mobility, self-care, usual activities, pain/discomfort and anxiety/depression of participants. This includes the EQ VAS, recording self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

REFERENCES:
- [Background] Chan EY, Phang KN, Glass GF Jr, Lim WS. Crossing, Trudging and Settling: A phenomenological inquiry into lived experience of Asian family caregivers of older persons with dementia. Geriatr Nurs. 2019 Sep-Oct;40(5):502-509. doi: 10.1016/j.gerinurse.2019.03.015. Epub 2019 Apr 9. PMID 30979516
- [Background] Sarafian V, Dimova P, Georgiev I, Taskov H. ABH blood group antigen significance as markers of endothelial differentiation of mesenchymal cells. Folia Med (Plovdiv). 1997;39(2):5-9. PMID 9314660
- [Background] Beynel P, Guigay J, Vauterin G. [Chronic cor pulmonale after embolism, antiphospholipid syndrome, Horton disease: therapeutic approach apropos of a case]. Rev Pneumol Clin. 1997;53(3):162-6. French. PMID 9296119
- [Background] Loke SXY, Chew EYH, Siew AL, Glass GF Jr, Chan EY. Transiting Back Home: Caregivers' Lived Experiences in Caring for Loved Ones on the Nasogastric Tube in the Home-Setting in Singapore. J Transcult Nurs. 2023 Sep;34(5):343-355. doi: 10.1177/10436596231175163. Epub 2023 May 24. PMID 37226459
- [Background] Saleh ZM, Williams GA, Taylor PC. Nuclear-magnetic-resonance relaxation in glassy Cu-As-Se and Cu-As-S. Phys Rev B Condens Matter. 1993 Mar 1;47(9):4990-5001. doi: 10.1103/physrevb.47.4990. No abstract available. PMID 10006659
- [Background] Coyle BR, Ubel PA. Spiritual values in the setting of health care priorities. Kennedy Inst Ethics J. 2000 Mar;10(1):107-8. No abstract available. PMID 11658152
- [Background] Leder SB. Serial fiberoptic endoscopic swallowing evaluations in the management of patients with dysphagia. Arch Phys Med Rehabil. 1998 Oct;79(10):1264-9. doi: 10.1016/s0003-9993(98)90273-8. PMID 9779682
- [Background] Garcia-Martinez J, Linares A, Suarez MD, Garcia-Peregrin E. [Effect of sulfhydryl reagents on mevalonate kinase partially purified from chicken liver]. Rev Esp Fisiol. 1982 Dec;38(4):393-6. Spanish. PMID 6302747